CLINICAL TRIAL: NCT07025512
Title: 177Lu-PSMA-617 in Metastatic Castration Resistant Prostate Cancer (mCRPC) With Bone Marrow Involvement and Cytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1690; NCI-2025-04173 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-06-06; First posted 2025-06-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Castration Resistant Prostate Cancer; Cytopenia; Anemia; Thrombocytopenia
MeSH Terms: conditions — Cytopenia; Anemia; Thrombocytopenia | interventions — Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SingleArm (Experimental): Treatment with 177Lu-PSMA-617
  Interventions: Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Given by IV

SUMMARY:
The purpose of the study is to examine the clinical and biological effects of 177Lu-PSMA-617 in mCRPC patients with cytopenia[s].

ELIGIBILITY:
Eligibility Criteria

1. Signed informed consent must be obtained before participation in the study. Participant subjects must be willing and able to provide consent.
2. Participants must be adults ≥18 years of age.
3. Histologically or cytologically confirmed adenocarcinoma of the prostate
4. Metastatic, castration-resistant prostate cancer (mCRPC) with a rise in PSA over a previous reference value measure 1 week prior. Minimal start value is 2.0 ng/mL
5. Has received ≥1 line prior systemic therapy approved in the metastatic and/or castrationresistant setting (in addition to androgen deprivation therapy [ADT])
6. Cytopenia due to prostate cancer involvement of bone marrow as documented by the presence of cancer cells in the BM sample and at least one of the below:

   1. Hemoglobin ≥7 g/dl and < 9 g/dl
   2. Pretransfusion Hemoglobin < 8 g/dl within 28 days for enrollment
   3. Platelet count ≥50 X 10 /L and ≤100 X 109 /L
7. Participants must agree to blood, bone marrow aspiration and biopsy collections at the specified time points.
8. Have had either orchiectomy OR be on luteinizing hormone-releasing hormone (LHRH) agonist or antagonist therapy with serum testosterone <50 ng/dL AND agree to stay on LHRH agonist or antagonist therapy during the study.
9. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
10. Serum creatinine ≤1.5 x ULN or estimated glomerular filtration rate >50 mL/min.
11. Adequate hepatic function:

    1. Total bilirubin ≤1.5 x ULN (≤3 x ULN if tumor liver involvement)
    2. AST ≤2.5 x ULN (≤5 x ULN if tumor liver involvement)
    3. ALT ≤2.5 x ULN (≤5 x ULN if tumor liver involvement)
12. Participants must have a positive 68Ga-PSMA-11 PET/CT scan, defined by at least 1 PSMA positive lesion with uptake > liver parenchyma in one or more metastatic lesions of any size in any organ system.
13. To avoid the risk of drug exposure through the ejaculate (even men with vasectomies), subjects must use a condom during sexual activity while on the study drug and for 6 months following the last dose of the study drug. If the subject is engaged in sexual activity with a woman of childbearing potential, a condom is required along with another effective contraceptive method consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies and their partners. Donation of sperm is not allowed while on the study drug and for 6 months following the last dose of the study drug.

Exclusion Criteria

1. Has primary bone marrow disorder (e.g. leukemia, myeloproliferative or myelodysplastic disorder)
2. Presence of iron deficiency or other hematological disorders that may cause anemia and cytopenia
3. Has participated in a study of an investigational agent or an investigational device within 4 weeks of the first dose of study therapy
4. Has received treatment with an approved systemic therapy within 2 weeks of dosing or has not yet recovered (i.e., grade ≤1 or baseline) from any acute toxicities attributed to the systemic therapy.
5. Has received radiation therapy or major surgery within 14 days of first administration of study drug.
6. Has received radiopharmaceutical agents in the past (e.g., Strontium-89, PSMA-targeted radioligand therapy)
7. Has received prior PSMA-targeting therapy
8. Another malignancy that is progressing or requires active treatment with the exception of non-melanoma skin cancer that has undergone potentially curative therapy
9. Untreated or active primary brain tumor, CNS metastases, leptomeningeal disease, or spinal cord compression
10. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection; or diagnosis of immunodeficiency
11. Has known allergy or hypersensitivity to study drugs
12. Concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, Poly Adenosine Diphosphate-Ribose Polymerase (PARP) inhibitor, biological therapy, or investigational or anti-cancer therapy
13. Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, uncontrolled infection, known active hepatitis B or C, or other significant co-morbid conditions that, in the opinion of the investigator, would impair study participation or cooperation
14. No active clinically significant cardiac disease is defined as any of the following:

    a. History or current diagnosis of ECG abnormalities indicating a significant risk of safety for participants in the study, such as i. Concomitant clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia, complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bi-fascicular block, Mobitz type II and third-degree AV block) ii. History of familial long QT syndrome or known family history of Torsades de Pointes
15. History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study
16. Symptomatic cord compression, unstable vertebral metastasis or clinical or radiologic findings indicative of impending cord compression

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 40 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs). | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Bagi Jana, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org